CLINICAL TRIAL: NCT03682770
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Study in Pediatric Subjects With Peanut Allergy to Evaluate the Efficacy and Safety of Dupilumab as Adjunct to AR101 (Peanut Oral Immunotherapy)
Brief Title: Study in Pediatric Subjects With Peanut Allergy to Evaluate Efficacy and Safety of Dupilumab as Adjunct to AR101 (Peanut Oral Immunotherapy)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry); Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-ALG-16114
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dupilumab + AR101 (Experimental): Participant randomization of a ratio of 2 active dupilumab arms
  Interventions: Drug: Dupilumab; Drug: AR101
- placebo matching dupilumab + AR101 (Experimental): Participant randomization of a ratio of 1 placebo arm
  Interventions: Drug: Placebo matching dupilumab; Drug: AR101

INTERVENTIONS:
Drug: Dupilumab — Dupilumab will be administered subcutaneously (SC) in a single-use, pre-filled glass syringe every two weeks (Q2W)
  Arms: dupilumab + AR101
Drug: Placebo matching dupilumab — Placebo matching dupilumab is prepared in the same formulation without the addition of protein
  Arms: placebo matching dupilumab + AR101
Drug: AR101 — AR101 will be provided in dose-escalating capsules and then sachets during maintenance phase

SUMMARY:
Primary objective is to assess whether dupilumab as adjunct to AR101 compared to placebo improves desensitization at the completion of up-dosing, defined as an increase in the proportion of participants who pass a post up-dosing double-blind placebo-controlled food challenge (DBPCFC) at visit 16.

Secondary objectives are:

* To assess whether dupilumab as adjunct to AR101 compared to placebo improves desensitization at the completion of up-dosing, defined as an increase in the cumulative tolerated dose (log transformed) of peanut protein during a post up-dosing DBPCFC at visit 16
* To assess whether dupilumab as (indefinite [continuously]) adjunct to AR101 compared to placebo maintains desensitization, defined as an increase in the proportion of participants who pass a post maintenance DBPCFC at visit 22
* To assess whether dupilumab as (limited [previously]) adjunct to AR101 compared to placebo maintains desensitization, defined as an increase in the proportion of participants who pass a post maintenance DBPCFC at visit 22
* To evaluate the safety and tolerability of dupilumab as adjunct to AR101 compared to placebo
* To assess the effect of dupilumab (compared to placebo) as adjunct to AR101 on the change in peanut-specific Immunoglobulin E (sIgE), Immunoglobulin G (IgG), Immunoglobulin G4 (IgG4), and peanut-specific IgG4/IgE ratio
* To assess if dupilumab increases the tolerability of AR101 as measured by the daily symptoms (electronic diary [e-diary]) during the up-dosing phase

ELIGIBILITY:
Key Inclusion Criteria:

* Experience dose-limiting symptoms at or before the challenge dose of peanut protein on screening and not experiencing dose-limiting symptoms to placebo as defined in the protocol
* Serum Immunoglobulin E (IgE) to peanut of ≥10 kUA/L and/or a skin prick test (SPT) to peanut ≥8 mm compared to a negative control
* Participants/legal guardians must be trained on the proper use of the epinephrine autoinjector device to be allowed to enroll in the study
* Participants with other known food allergies must agree to eliminate these other food items from their diet so as not to confound the safety and efficacy data from the study

Key Exclusion Criteria:

* History of other chronic disease (other than asthma, Atopic Dermatitis (AD), or allergic rhinitis) requiring therapy (eg, heart disease, diabetes, hypertension) that would represent a risk to participant's health or safety in this study or ability to comply with study protocol
* History of frequent or recent severe, life-threatening episode of anaphylaxis or anaphylactic shock
* History of eosinophilic Gastrointestinal (GI) disease
* Asthma at time of enrollment with any of the following:

  * Forced Expiratory Volume 1 Second (FEV1) <80% of predicted or ratio of FEV1 to forced vital capacity (FEV1/FVC) <75% of predicted with or without controller medications
  * Inhaled corticosteroids (ICS) dosing of daily fluticasone (or equivalent ICS based on NHLBI dosing chart)
  * One hospitalization in the past year for asthma
  * Emergency room visit for asthma within 6 months prior to screening
* Use of systemic corticosteroids within 2 months prior to screening
* Use of other forms of allergen immunotherapy or immunomodulatory therapy within 3 months prior to screening
* Use of any agents known or likely to interact with epinephrine (eg, beta-blockers, angiotensin converting enzyme-inhibitors, tri-cyclic antidepressants, or other drugs), within 3 weeks prior to screening
* Allergy to oat (placebo in DBPCFC)

Note: Other protocol Inclusion/Exclusion Criteria apply

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (24):
- United States (24):
  - Regeneron Investigational Site, Birmingham, Alabama
  - Regeneron Investigational Site, Tucson, Arizona
  - Regeneron Investigational Site, Little Rock, Arkansas
  - Regeneron Investigational Site, Los Angeles, California
  - Regeneron Investigational Site, Mission Viejo, California
  - Regeneron Investigational Site, Mountain View, California
  - Regeneron Investigational Site, Rolling Hills Estates, California
  - Regeneron Investigational Site, Denver, Colorado
  - Regeneron Investigational Site, Washington D.C., District of Columbia
  - Regeneron Investigational Site, Tampa, Florida
  - Regeneron Investigational Site, Atlanta, Georgia
  - Regeneron Investigational Site, Marietta, Georgia
  - Regeneron Investigational Site, Chicago, Illinois
  - Regeneron Investigational Site, Baltimore, Maryland
  - Regeneron Investigational Site, Boston, Massachusetts
  - Regeneron Investigational Site, Ann Arbor, Michigan
  - Regeneron Investigational Site, Ypsilanti, Michigan
  - Regeneron Investigational Site, Minneapolis, Minnesota
  - Regeneron Investigational Site, Ocean Township, New Jersey
  - Regeneron Investigational Site, Great Neck, New York
  - Regeneron Investigational Site, New York, New York
  - Regeneron Investigational Site, Chapel Hill, North Carolina
  - Regeneron Investigational Site, Philadelphia, Pennsylvania
  - Regeneron Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] Ghelli C, Costanzo G, Canonica GW, Heffler E, Paoletti G. New evidence in food allergies treatment. Curr Opin Allergy Clin Immunol. 2024 Aug 1;24(4):251-256. doi: 10.1097/ACI.0000000000000999. Epub 2024 May 30. PMID 38814736

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 232 participants were screened; 148 participants were randomized. Of the 84 not randomized, 53 did not meet inclusion/exclusion criteria and 13 withdrew consent.
Groups:
- Pre-AR101 Dosing Period: Placebo-matched Dupilumab: Participants received placebo-matched dupilumab
- Pre-AR101 Dosing Period: Dupilumab: Participants of ≥60 kilograms (kg) body weight (BW) received dupilumab 300 milligrams (mg) subcutaneously (SC) every 2 weeks (Q2W); participants of ≥ 30kg to < 60kg BW received dupilumab 200 mg SC Q2W; participants of <30kg BW received dupilumab 100 mg SC Q2W
- AR101 Up-dosing Period: Placebo + AR101: Participants who received placebo-matched dupilumab in the pre-AR101 dosing period received placebo in combination with a gradual up-dosing of AR101 oral capsules
- AR101 Up-dosing Period: Dupilumab + AR101: Participants who received dupilumab in the pre-AR101 dosing period received dupilumab during the up-dosing period in combination with a gradual up-dosing of AR101 oral capsules
- AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued: Participants who received placebo-matched dupilumab + AR101 in the up-dosing period continued in the maintenance period
- AR101 Maintenance Period: Dupilumab + AR101 Continued: Participants who received dupilumab + AR101 in up-dosing period continued to receive dupilumab + AR101 in the maintenance period
- AR101 Maintenance Period: Dupilumab + AR101/Placebo-matched Dupilumab + AR101: Participants who received dupilumab + AR101 in the up-dosing period switched to placebo-matched dupilumab + AR101 in the maintenance period
Period: Pre-AR101 Dosing Period (Day 1 - Week 4)
Arm/Group | Pre-AR101 Dosing Period: Placebo-matched Dupilumab | Pre-AR101 Dosing Period: Dupilumab | AR101 Up-dosing Period: Placebo + AR101 | AR101 Up-dosing Period: Dupilumab + AR101 | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101/Placebo-matched Dupilumab + AR101
Started | 50 | 98 | 0 | 0 | 0 | 0 | 0
Completed (Completed = Progressed to Up-dosing period) | 49 | 96 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor decision | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: AR101 Up-dosing Period (Week 28-40)
Arm/Group | Pre-AR101 Dosing Period: Placebo-matched Dupilumab | Pre-AR101 Dosing Period: Dupilumab | AR101 Up-dosing Period: Placebo + AR101 | AR101 Up-dosing Period: Dupilumab + AR101 | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101/Placebo-matched Dupilumab + AR101
Started | 0 | 0 | 49 | 96 | 0 | 0 | 0
Completed (Completed = Progressed to Maintenance period) | 0 | 0 | 39 | 88 | 0 | 0 | 0
Not Completed | 0 | 0 | 10 | 8 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 3 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Investigator/Sponsor decision | 0 | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Chronic/recurrent GI AEs/Symptoms | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 2 | 0 | 0 | 0
Period: AR101 Maintenance Period: (Week 52-64)
Arm/Group | Pre-AR101 Dosing Period: Placebo-matched Dupilumab | Pre-AR101 Dosing Period: Dupilumab | AR101 Up-dosing Period: Placebo + AR101 | AR101 Up-dosing Period: Dupilumab + AR101 | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101/Placebo-matched Dupilumab + AR101
Started (Randomized) | 0 | 0 | 0 | 0 | 40 (Participants who completed and ongoing in Up-dosing Period: placebo + AR101 were randomized into the AR101 maintenance period. One additional participant was randomized and received treatment in placebo + AR101 group in AR101 maintenance period.) | 44 (Participants who completed and ongoing in Up-dosing Period: dupilumab + AR101 were re-randomized (1:1) ratio into the AR101 maintenance period.) | 44 (Participants who completed and ongoing in Up-dosing Period: dupilumab + AR101 were re-randomized (1:1) ratio into the AR101 maintenance period.)
Randomized and Treated | 0 | 0 | 0 | 0 | 40 | 43 | 42
Completed | 0 | 0 | 0 | 0 | 36 | 41 | 41
Not Completed | 0 | 0 | 0 | 0 | 4 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 1 | 1
Not completed — Investigator/Sponsor decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Randomized, but not treated | 0 | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-AR101 Dosing Period: Placebo-matched Dupilumab | Pre-AR101 Dosing Period: Dupilumab | Total
Number analyzed (Participants) | 50 | 98 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (3.00) | 11.3 (3.12) | 11.1 (3.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 38 | 56
  Male | 32 | 60 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 45 | 87 | 132
  Unknown or Not Reported | 1 | 3 | 4
Race/Ethnicity, Customized [Number; unit: participants] — Race
  participants
    White | 40 | 70 | 110
    Black or African American | 1 | 3 | 4
    Asian | 7 | 18 | 25
    American Indian or Alaska Native | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Other | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Treated With Dupilumab Plus AR101 vs Placebo Plus AR101 Who Passed a Post Up-dosing Double-blind, Placebo-controlled Food Challenge (DBPCFC) With 2044 mg (Cumulative) Peanut Protein at Visit 16 (Week 28 to 40)
Description: Symptoms considered to be allergic were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions. The allergic reaction is measured on a 1-5 scale, with grade 1 being mild, grade 2 being moderate, grade 3 being severe, grade 4 being life threatening, and grade 5 as death. the higher the grade, the more severe the allergic reaction. Participants were considered to have passed the DBPCFC if they did not experience any objective Grade 1 reaction. Percentage of participants treated with dupilumab plus AR101 vs placebo plus AR101 who passed a post up-dosing DBPCFC with 2044 mg (Cumulative) peanut protein at Visit 16 (Week 28 to 40) was reported. Cumulative data during the specified period was calculated as the average of all available post-randomization values during the specified time period (Week 28 to Week 40).
Time Frame: At Visit 16 (Week 28 to 40)
Population: Modified full analysis set (mFAS) included all participants in the full analysis set (FAS) who underwent biweekly in-clinic up-dosing as described/specified in the protocol and underwent the post up-dosing DBPCFC at Visit 16 (Weeks 28 to 40). Data were planned to be reported and analyzed only for AR101 Up-dosing Period: Dupilumab plus AR101 vs Placebo plus AR101.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AR101 Up-dosing Period: Placebo + AR101 | AR101 Up-dosing Period: Dupilumab + AR101
Number analyzed (Participants) | 39 | 84
Percentage of participants | 35.90 [21.204 to 52.820] | 55.95 [44.695 to 66.778]
Statistical Analysis 1: Comparison: AR101 Up-dosing Period: Placebo + AR101 vs AR101 Up-dosing Period: Dupilumab + AR101; Test type: Superiority; p = 0.0420, Cochran-Mantel-Haenszel — The p-value was derived by Cochran-Mantel-Haenszel (CMH) test stratified by screening peanut-specific IgE level and baseline body weight; Difference in percentage = 20.23, 95% CI 2-sided [1.266 to 39.189] — Difference in percentage derived by Mantel-Haenszel (MH) method

2. Secondary Outcome: Change From Baseline in Cumulative Tolerated Dose (Log Transformed) of Peanut Protein During a DBPCFC at Visit 16 (Week 28 to 40) in Participants Treated With Dupilumab Plus AR101 vs Placebo Plus AR101
Description: Change from baseline in cumulative tolerated dose (log transformed) of peanut protein during a DBPCFC at Visit 16 (Week 28 to 40) in participants treated with dupilumab plus AR101 vs placebo plus AR101 was reported. Cumulative tolerated dose during the specified period was calculated as the mean of all available post-randomization values during the specified time period (Week 28 to Week 40).
Time Frame: Baseline, Visit 16 (Week 28 to 40)
Population: mFAS included all participants in the FAS who underwent biweekly in-clinic up-dosing as described/specified in the protocol and underwent the post up-dosing DBPCFC at Visit 16 (Weeks 28 to 40). Data were planned to be reported and analyzed only for AR101 Up-dosing Period: Dupilumab plus AR101 vs Placebo plus AR101.
Measure: Least Squares Mean (Standard Error); unit: Log Transformed Milligrams
Arm/Group | AR101 Up-dosing Period: Placebo + AR101 | AR101 Up-dosing Period: Dupilumab + AR101
Number analyzed (Participants) | 39 | 84
Log Transformed Milligrams | 3.78 (0.270) | 4.45 (0.205)
Statistical Analysis 1: Comparison: AR101 Up-dosing Period: Placebo + AR101 vs AR101 Up-dosing Period: Dupilumab + AR101; Test type: Superiority; p = 0.0400, ANCOVA — P-value is based on treatment difference (dupilumab + AR101 vs placebo + AR101) of the LS mean change using analysis of covariance (ANCOVA) model; Least Square Mean Difference = 0.67, 95% CI 2-sided [0.031 to 1.305]

3. Secondary Outcome: Percentage of Participants Treated With Dupilumab Plus AR101 vs Placebo Plus AR101 Who Reached the 300 mg/Day Dose of AR101 by Visit 16 (Week 28 to 40)
Description: Percentage of participants treated with dupilumab plus AR101 vs placebo plus AR101 who reached the 300 mg/day dose of AR101 by Visit 16 (Week 28 to 40) was reported. Cumulative data during the specified period was calculated as the average of all available post-randomization values during the specified time period (Week 28 to Week 40).
Time Frame: At Visit 16 (Week 28 to 40)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AR101 Up-dosing Period: Placebo + AR101 | AR101 Up-dosing Period: Dupilumab + AR101
Number analyzed (Participants) | 39 | 84
Percentage of participants | 76.92 [60.674 to 88.866] | 89.29 [80.633 to 94.982]
Statistical Analysis 1: Comparison: AR101 Up-dosing Period: Placebo + AR101 vs AR101 Up-dosing Period: Dupilumab + AR101; Test type: Superiority; p = 0.0806, Cochran-Mantel-Haenszel — P-values were derived by CMH test stratified by screening peanut-specific IgE level (<=100 kilo allergy unit per liter [kUA/L] vs >100 kUA/L) and body weight (<30 kg, >=30 and <60 kg, or >=60 kg); Difference in percentage = 11.91, 95% CI 2-sided [-3.612 to 27.440] — Difference in percentage derived by MH method

4. Secondary Outcome: Time From Randomization to the First Time When Participants Reached the 300 mg/Day Dose of AR101 During the Up-dosing Treatment Phase by Visit 16 (Week 28 to 40)
Description: Time (in days) from randomization to the first time when participants reached the 300 mg/day dose of AR101 during the up-dosing treatment phase by Visit 16 (Week 28 to 40) was reported. If participants did not reach the 300 mg/day dose of AR101 during the 28-week treatment period, they were censored at the date of their last visit during pre-AR101 dosing and AR101 up-dosing treatment period. Analysis was performed using Kaplan-Meier Estimated method.
Time Frame: At Visit 16 (Week 28 to 40)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AR101 Up-dosing Period: Placebo + AR101 | AR101 Up-dosing Period: Dupilumab + AR101
Number analyzed (Participants) | 39 | 84
Days | 164.6 (38.43) | 167.5 (32.01)

5. Secondary Outcome: Percentage of Participants (Continuously) Treated With Dupilumab Plus AR101 vs Placebo Plus AR101 Who Passed a Post Maintenance DBPCFC With 2044 mg (Cumulative) Peanut Protein at Visit 22 (Week 52 to 64)
Description: Symptoms considered to be allergic were graded using the CoFAR Grading Scale for Systemic Allergic Reactions. The allergic reaction is measured on a 1-5 scale, with grade 1 being mild, grade 2 being moderate, grade 3 being severe, grade 4 being life threatening, and grade 5 as death. the higher the grade, the more severe the allergic reaction. Participants were considered to have passed the DBPCFC if they did not experience any objective Grade 1 reaction. Percentage of participants (continuously) treated with dupilumab plus AR101 vs placebo plus AR101 who passed a post maintenance DBPCFC with 2044 mg (cumulative) peanut protein at Visit 22 (Week 52 to 64) was reported. Cumulative data during the specified period was calculated as the average of all available post-randomization values during the specified time period (Week 52 to Week 64).
Time Frame: At Visit 22 (Week 52 to 64)
Population: FAS-maintenance (a subset of FAS) included participants in the FAS who achieved 300 mg/day AR101 for at least 2 weeks in the up-dosing phase and re-randomized based on the treatment allocated by the IWRS at Visit 16 (Weeks 28 to 40). Data were planned to be reported and analyzed only for AR101 Maintenance Period: Continuously on Dupilumab plus AR101 vs Placebo plus AR101.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101 Continued
Number analyzed (Participants) | 40 | 44
Percentage of participants | 47.50 [31.512 to 63.872] | 56.82 [41.034 to 71.651]
Statistical Analysis 1: Comparison: AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued vs AR101 Maintenance Period: Dupilumab + AR101 Continued; Test type: Superiority; p = 0.3530, Cochran-Mantel-Haenszel — P-values were derived by CMH test stratified by screening peanut-specific IgE level (<=100 kUA/L vs >100 kUA/L) and baseline body weight (<30 kg, >=30 kg and <60 kg, or >=60 kg); Difference in percentage = 10.40, 95% CI 2-sided [-11.668 to 32.474] — Difference in percentage derived by MH method

6. Secondary Outcome: Change From Baseline in Cumulative Tolerated Dose (Log Transformed) of Peanut Protein During a DBPCFC at Visit 22 (Week 52 to 64) in Participants (Continuously) Treated With Dupilumab Plus AR101 vs Placebo Plus AR101
Description: Change from baseline in cumulative tolerated dose (log transformed) of peanut protein during a DBPCFC at Visit 22 (Week 52 to 64) in participants (continuously) treated with dupilumab plus AR101 vs placebo plus AR101 was reported. Cumulative tolerated dose during the specified period was calculated as the mean of all available post-randomization values during the specified time period (Week 52 to Week 64).
Time Frame: Baseline, Visit 22 (Week 52 to 64)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Log Transformed Milligrams
Arm/Group | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101 Continued
Number analyzed (Participants) | 40 | 44
Log Transformed Milligrams | 4.19 (0.245) | 4.56 (0.250)
Statistical Analysis 1: Comparison: AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued vs AR101 Maintenance Period: Dupilumab + AR101 Continued; Test type: Superiority; p = 0.2628, ANCOVA — P-value is based on treatment difference of the LS mean change using ANCOVA model with baseline tolerated cumulative amount of peanut protein DBPCFC (log transformed) as covariate and the treatment screening peanut-specific IgE level and baseline; Least Square Mean Difference = 0.37, 95% CI 2-sided [-0.281 to 1.029]

7. Secondary Outcome: Percentage of Participants (Previously) Treated With Dupilumab + AR101/Placebo +AR101 vs Placebo Plus AR101 Who Passed a Post Maintenance DBPCFC With 2044 mg (Cumulative) Peanut Protein at Visit 22 (Week 52 to 64)
Description: Symptoms considered to be allergic were graded using the CoFAR Grading Scale for Systemic Allergic Reactions. The allergic reaction is measured on a 1-5 scale, with grade 1 being mild, grade 2 being moderate, grade 3 being severe, grade 4 being life threatening, and grade 5 as death. the higher the grade, the more severe the allergic reaction. Participants were considered to have passed the DBPCFC if they did not experience any objective Grade 1 reaction. Percentage of participants (previously) treated with dupilumab plus AR101 (and re-randomized to placebo plus AR101) vs placebo plus AR101 who "pass" a post maintenance DBPCFC with 2044 mg (cumulative) peanut protein at Visit 22 (Week 52 to 64) was reported. Cumulative data during the specified period was calculated as the average of all available post-randomization values during the specified time period (Week 52 to Week 64).
Time Frame: At Visit 22 (Week 52 to 64)
Population: FAS-maintenance (a subset of FAS) included participants in the FAS who achieved 300 mg/day AR101 for at least 2 weeks in the up-dosing phase and re-randomized based on the treatment allocated by the IWRS at Visit 16 (Weeks 28 to 40). Data were planned to be reported and analyzed only for AR101 Maintenance Period: Dupilumab + AR101/Placebo +AR101 vs Placebo + AR101.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101/Placebo-matched Dupilumab + AR101
Number analyzed (Participants) | 40 | 44
Percentage of participants | 47.50 [31.512 to 63.872] | 45.45 [30.391 to 61.153]
Statistical Analysis 1: Comparison: AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued vs AR101 Maintenance Period: Dupilumab + AR101/Placebo-matched Dupilumab + AR101; Test type: Superiority; p = 0.8140, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]; Difference in percentage = -2.36, 95% CI 2-sided [-25.004 to 20.282] — Difference in percentage derived by MH method

8. Secondary Outcome: Change From Baseline in Cumulative Tolerated Dose (Log Transformed) of Peanut Protein During a DBPCFC at Visit 22 (Week 52 to 64) in Participants (Previously) Treated With Dupilumab + AR101/Placebo +AR101 vs Placebo Plus AR101
Description: Change from baseline in cumulative tolerated dose (log transformed) of peanut protein during a DBPCFC at Visit 22 (Week 52 to 64) in participants (previously) treated with dupilumab plus AR101 (and re-randomized to placebo plus AR101) vs placebo plus AR101 was reported. Cumulative tolerated dose during the specified period was calculated as the mean of all available post-randomization values during the specified time period (Week 52 to Week 64).
Time Frame: Baseline, Visit 22 (Week 52 to 64)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Log Transformed Milligrams
Arm/Group | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101/Placebo-matched Dupilumab + AR101
Number analyzed (Participants) | 40 | 44
Log Transformed Milligrams | 4.19 (0.245) | 4.14 (0.244)
Statistical Analysis 1: Comparison: AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued vs AR101 Maintenance Period: Dupilumab + AR101/Placebo-matched Dupilumab + AR101; Test type: Superiority; p = 0.8805, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Square Mean Difference = -0.05, 95% CI 2-sided [-0.699 to 0.599]

9. Secondary Outcome: Percent Change From Baseline in Peanut-specific IgE in Participants Treated With Dupilumab Plus AR101 vs Placebo Plus AR101 to Visit 16 (Week 28 to 40)
Description: Percent change from baseline in peanut-specific IgE in participants treated with dupilumab + AR101 vs placebo + AR101 to Visit 16 (Week 28 to 40) was reported. Analysis was performed using Last observation carried forward (LOCF) method. Data reported during the specified period was calculated as the average of all available post-randomization values during the specified time period (Week 28 to Week 40).
Time Frame: Baseline up to Visit 16 (Weeks 28 to 40)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | AR101 Up-dosing Period: Placebo + AR101 | AR101 Up-dosing Period: Dupilumab + AR101
Number analyzed (Participants) | 39 | 84
Percent change | 29.9 [3.3 to 82.2] | -60.6 [-68.1 to -50.5]

10. Secondary Outcome: Percent Change From Baseline in Peanut-specific IgE in Participants (Continuously) Treated With Dupilumab Plus AR101 vs Placebo Plus AR101 to Visit 22 (Week 52 to 64)
Description: Percent change from baseline in peanut-specific IgE in participants treated with dupilumab + AR101 vs placebo + AR101 to Visit 22 (Week 52 to 64) was reported. Analysis was performed using LOCF method. Data reported during the specified period was calculated as the average of all available post-randomization values during the specified time period (Week 52 to Week 64).
Time Frame: Baseline up to Visit 22 (Week 52 to 64)
Population: mFAS-maintenance (a subset of mFAS) included participants in the mFAS who achieved 300 mg/day AR101 for at-least 2 weeks in the up-dosing phase and re-randomized based on the treatment allocated by the IWRS at Visit 16 (Weeks 28 to 40). Data were planned to be reported and analyzed only for AR101 Maintenance Period: Continuously on Dupilumab Plus AR101 vs Placebo Plus AR101.
Measure: Median (Full Range); unit: Percent change
Arm/Group | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101 Continued
Number analyzed (Participants) | 29 | 36
Percent change | 10.1 [-73.3 to 98.5] | -73.7 [-91.7 to -52.5]
Statistical Analysis 1: Comparison: AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued vs AR101 Maintenance Period: Dupilumab + AR101 Continued; Test type: Superiority; p < 0.0001, ANCOVA — P-value was based on treatment difference (vs. Continuously on Placebo + AR101) in percent change from baseline using rank-based ANCOVA model with baseline measurement as covariate,- and stratification factors and the treatment as fixed factors; Difference percentage = -85.55, 95% CI 2-sided [-99.47 to -73.91] — Median difference and its 95% CIs were estimated with the Hodges-Lehmann method

11. Secondary Outcome: Percent Change From Baseline in Peanut-specific IgE in Participants (Continuously) Treated With Dupilumab Plus AR101 vs Placebo Plus AR101 to Visit 25 (Weeks 64 to 76)
Description: Percent change from baseline in peanut-specific IgE in participants treated with dupilumab + AR101 vs placebo + AR101 to Visit 25 (Week 64 to 76) was reported. Analysis was performed using LOCF method. Data reported during the specified period was calculated as the average of all available post-randomization values during the specified time period (Week 64 to Week 76).
Time Frame: Baseline up to Visit 25 (Weeks 64 to 76)
Population: as for outcome 10
Measure: Median (Full Range); unit: Percent change
Arm/Group | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101 Continued
Number analyzed (Participants) | 29 | 36
Percent change | -7.2 [-84.6 to 94.7] | -73.9 [-91.6 to -45.5]
Statistical Analysis 1: Comparison: AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued vs AR101 Maintenance Period: Dupilumab + AR101 Continued; Test type: Superiority; p < 0.0001, ANCOVA — P-value was based on treatment difference (vs. Continuously on Placebo + AR101) in percent change from baseline using rank-based ANCOVA model with baseline measurement as covariate, and stratification factors and the treatment as fixed factors; Difference in percentage = -68.78, 95% CI 2-sided [-86.71 to -56.40] — Median difference and its 95% CIs were estimated with the Hodges-Lehmann method

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 76
Arm/Group | Pre-AR101 Dosing Period: Placebo-matched Dupilumab | Pre-AR101 Dosing Period: Dupilumab | AR101 Up-dosing Period: Placebo + AR101 | AR101 Up-dosing Period: Dupilumab + AR101 | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101 Continued | AR101 Maintenance Period: Dupilumab + AR101/Placebo-matched Dupilumab + AR101
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/98 | 0/49 | 0/96 | 0/40 | 0/42 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/98 | 0/49 | 0/96 | 0/40 | 1/42 | 0/43
Other Adverse Events (participants affected / at risk) | 12/50 | 23/98 | 34/49 | 47/96 | 13/40 | 17/42 | 15/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-AR101 Dosing Period: Placebo-matched Dupilumab (N=50) | Pre-AR101 Dosing Period: Dupilumab (N=98) | AR101 Up-dosing Period: Placebo + AR101 (N=49) | AR101 Up-dosing Period: Dupilumab + AR101 (N=96) | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued (N=40) | AR101 Maintenance Period: Dupilumab + AR101 Continued (N=42) | AR101 Maintenance Period: Dupilumab + AR101/Placebo-matched Dupilumab + AR101 (N=43)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-AR101 Dosing Period: Placebo-matched Dupilumab (N=50) | Pre-AR101 Dosing Period: Dupilumab (N=98) | AR101 Up-dosing Period: Placebo + AR101 (N=49) | AR101 Up-dosing Period: Dupilumab + AR101 (N=96) | AR101 Maintenance Period: Placebo-matched Dupilumab + AR101 Continued (N=40) | AR101 Maintenance Period: Dupilumab + AR101 Continued (N=42) | AR101 Maintenance Period: Dupilumab + AR101/Placebo-matched Dupilumab + AR101 (N=43)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2) | 7 (9) | 16 (21) | 1 (2) | 5 (8) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 7 (13) | 0 (0) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (10) | 9 (12) | 1 (1) | 4 (9) | 3 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (5) | 8 (12) | 1 (1) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (7) | 6 (7) | 0 (0) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 8 (11) | 5 (6) | 1 (1) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (6) | 5 (7) | 0 (0) | 3 (5) | 1 (2)
Oral pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4) | 4 (8) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 7 (11) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (6) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (7) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 5 (9) | 3 (13) | 6 (14) | 1 (2) | 1 (1) | 0 (0)
Injection site urticaria (General disorders) | 2 (2) | 5 (7) | 2 (9) | 5 (14) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 2 (2) | 5 (6) | 0 (0) | 2 (3) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (6) | 0 (0) | 3 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 1 (2) | 2 (2) | 3 (4)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 4 (8) | 5 (9) | 1 (6) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (6) | 3 (7) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 3 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT03682770/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03682770/SAP_001.pdf